CLINICAL TRIAL: NCT03839004
Title: "MYND&CO: Studio Pilota Sull'Evoluzione Della Salute Psico-fisica Della Donna in Gravidanza Secondo Una modalità Multidisciplinare e Personalizzata"
Brief Title: MYND&CO: Studio Pilota Dell'Evoluzione Della Salute Psico-fisica Della Donna in Gravidanza
Acronym: MYND&CO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MYND&CO
Record Dates: First submitted 2019-01-10; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Pregnancy; Mental Health Wellness 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 200 woman with single spontaneous pregnancies who recieve, as well as traditional obstetrical care, yoga classes, myndfulness classes, coaching, nutrition counselling and osteopathic treatment
  Interventions: Behavioral: Integrated approach to pregnancy
- Controls (No Intervention): 200 woman with single spontaneous pregnancies recieving traditional obstetrical care

INTERVENTIONS:
Behavioral: Integrated approach to pregnancy — Yoga classes, mindfulness classes, coaching, nutrition counselling and osteopathy
  Arms: Intervention group

SUMMARY:
To evaluate an integral approach to the maternal-fetal diad.

A randomized non farmacological monocentric trial.

400 women with single spontaneous pregnancies are randomized.

200 recieve standardized traditional obstetrical care

200 recieve nutritional advice, osteopathic treatment, yoga classes, mindfulness classes and coaching as well as regular obstetrical care.

We evaluate the psychological status at recruitment, at the end of pregnancy and 40 days after birth.

DETAILED DESCRIPTION:
The first international scientific research project focusing on a holistic approach to pregnancy is starting now at the Clinica Mangiagalli in Milan.

This innovative model aims to the gold standard of a "positive pregnancy", which supports both the somatic and psychological component of the mother-newborn unit, and thus organically and proactively prevents the main issues arising during pregnancy and delivery due to unhealthy lifestyles.

A team of experts will take comprehensive care of the mother, first by means of an accurate evaluation of her nutritional profile, and then of her biomechanic (osteo-skeletal) state.

Then, the experts will lead an "academic" path, which will initiate a development of her biochemistry (through nutrition), respiration (through yoga), physical wellbeing (through osteopathy and yoga); and strengthen her sense of self, removing her self-doubt (through mindfulness and yoga).

The women will be supported up until childbirth, so as to attempt to prevent the main complications of pregnancy and of delivery.

This model does not aim to substitute the allopathic one which is currently in place (ultrasounds, ob-gyn appointments, tests, etc.), but to enhance its nature in a more effectively THERAPEUTIC manner, increasing the mother-newborn unit's potential of health.

In summary:

* Weekly mindfulness meet-ups
* Weekly yoga meet-ups
* Nutritional screening and further check-ups, if needed
* Osteopathic screening
* Five motivational meetings with a coach
* Four obstetrical appointments
* Obstetrical screening and check-ups up until childbirth

The team in charge of the project is made up of gynaecologists, midwives, psychologists, osteopaths, nutritionists and yoga teachers, who all collaborate on a regular basis with the Clinica Mangiagalli.

The project is offered to women free of charge.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancies
* spontaneous pregnancies
* no maternal medical conditions
* no language barrier

Exclusion Criteria:

* maternal or fetal medical conditions
* age <18 or <45
* ivf
* language barrier
* multiple pregnancies

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 400 (Estimated)
Dates: Start 2019-01-08 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Evolution in women's mental health from t0( first trimester) to after birth (40 days after delivery) | from third month of pregnancy to 1 month after delivery
  evaluated by the means of psychological questionaire SF12
Woman's physical health during pregnancy | from first trimester of pregnancy to day of delivery
  weight gain in pregnancy
Diagnosis of pregnancy-related diabetes | from 24 weeks of pregnancy to the day of delivery
  positive blood glucose curve or fasting glucose >92 on 2 different measurements
Diagnosis of pregnancy-related hypertension | from the 20th week of gestation to 40 days after delivery
  diagnosis of hypertension from the 20th week of gestation to 40 days after delivery
Woman's osteo-muscular health during pregnancy | from the 20th week of gestation to 40 days after delivery
  diagnosis of low back pain and sciatic nerve pain during pregnancy
Quality of delivery | birth
  number of operative deliveries/ cesarean sections
Newborn's health | birth
  apgar
Newborn's pH | birth
  pH at birth
Newborn's weight | birth
  weight at birth
Newborn's blood gas | birth
  blood gas at birth

CONTACTS AND LOCATIONS:
Overall Officials: Niccolò Giovannini, MD, Principal Investigator — IRCCS Clinica Mangiagalli
Locations (1):
- Fondazione IRCCS Ca' Granda, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be shared

REFERENCES:
- [Derived] Giovannini N, Cetera GE, Ercolino C, Miozzo MR, Parazzini F, Ferrazzi EM, Manzotti A, Colaceci S. MYNd&CO (Mindfulness, Yoga, Nutrition, development & Coaching, and Osteopathy) randomized controlled trial for a positive psychophysical experience in pregnancy and after birth: a study protocol. Acta Biomed. 2021 Jul 29;92(S2):e2021032. doi: 10.23750/abm.v92iS2.11259. PMID 34328141